CLINICAL TRIAL: NCT02991872
Title: A Phase IV, Open Label, Single-center Extension Study, to Evaluate the Long-term Persistence of Immune Responses After Post-exposure Prophylaxis With Purified Chicken-embryo Cell Rabies Vaccine in Chinese Children
Brief Title: A Study to Evaluate Persistence of Immune Responses After Post-exposure Prophylaxis of Rabipur® (Purified Chicken-embryo Cell Rabies Vaccine) in Chinese Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 205634; V49_24E1 (Other: Novartis)
Record Dates: First submitted 2016-12-09; First posted 2016-12-14 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Virus Diseases
Keywords: Persistence; Purified chicken-embryo cell rabies vaccine; Rabies Virus Neutralizing Antibody (RVNA); Immunogenicity; Post-Exposure Prophylaxis (PEP); Rabipur
MeSH Terms: conditions — Virus Diseases | interventions — Blood Specimen Collection

ARMS (1):
- V49_24E1 Group (Other): Up to 225 subjects, who completed the full PEP rabies regimens in the parent study V49_24 (NCT01680016), will be invited to participate to this extension study.
  Interventions: Procedure: Blood draw

INTERVENTIONS:
Procedure: Blood draw — Subjects aged from ≥6 to ≤17 years at the time of enrolment in the parent clinical trial (following the CFDA post-marketing commitment requirement) and who received the full PEP rabies regimen as an intramuscular injection according to the vaccine group to which they were assigned in the V49_24 (NCT01680016) study will be invited to take part in this study. Single blood draw from subjects at Day-1/Visit-1. Subjects will be observed for 15 minutes after the blood draw.

SUMMARY:
The purpose of this study is to evaluate the long-term persistence of immune responses approximately 5 years or more after simulated rabies post-exposure prophylaxis provided in 2012 according to Essen (1-1-1-1-1) or Zagreb (2-1-1) intramuscular (IM) regimens in the subset of subjects who participated in the parent study (V49_24 [NCT01680016]) who were aged ≥6 and ≤17 years at the time of enrollment.

This study is aimed to respond to a post-marketing commitment by the China Food and Drug Administration (CFDA) requested at the time of the renewal of the purified chicken-embryo cell rabies vaccine license in China, granted in August 2015.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with age ≥ 6 and ≤17 at the time of enrollment in the parent study who signed the informed consent prior to the extension study entry, who received the full PEP in the parent study according to either the Zagreb or Essen intramuscular regimens.
2. Subjects who or whose parent(s)/legal guardian(s) have voluntarily given written informed consent/assent for this extension study after the nature of the study has been explained according to local regulatory requirements, prior to study entry.
3. Individuals who can comply with study procedures.

Exclusion Criteria:

Prior to extension study entry, each subject must not have:

1. Documented medical history of exposure to rabies or rabies prophylaxis after completion of the parent study (V49_24 [NCT01680016]) and before study start.
2. Participated in the parent study (V49_24 [NCT01680016]) but not received the full PEP vaccination course (or received it out of window) following assignment to either Zagreb or Essen regimen during the parent study.
3. Progressive, unstable or uncontrolled clinical conditions.
4. Clinical conditions representing a contraindication to blood draws.
5. Abnormal function of the immune system resulting from:

   1. Clinical conditions.
   2. Systemic administration of corticosteroids for more than 14 consecutive days within 90 days prior to informed consent for all age groups.
   3. Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to informed consent for all age groups.
6. Received immunoglobulins or any blood products within 180 days prior to informed consent for all age groups.
7. Study personnel as an immediate family or household member.
8. Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the subject due to participation in the study.

Ages: 10 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2017-03-12 (Actual); Study Completion 2017-03-12 (Actual)

PRIMARY OUTCOMES:
Rabies Virus Neutralizing Antibody(RVNA) GMCs as measured by rapid fluorescent focus inhibition test(RFFIT) measured in the study, following the Post-Exposure Prophylaxis(PEP) received in the V49_24 (NCT01680016) parent study (Zagreb and Essen regimens). | Day-1/Visit-1
Percentage of subjects with RVNA concentration ≥ 0.5 IU/mL measured in this study, following the PEP received in the V49_24 (NCT01680016) parent study (Zagreb and Essen regimens). | Day-1/Visit-1

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Mengshan, China